CLINICAL TRIAL: NCT05139537
Title: Association of Vestibular and Postural Impairments With Functional Status in Stroke
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Maryam Bashir
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: vestibular impairments, functional status.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
: Stroke is leading cause of long-term disability in individuals. The location and extent of brain injury determines the severity of neurological deficits. The incidence of stroke dramatically increases in old age. Patients with stroke always come across with problems associated with balance, vertigo, dizziness and posture resulting in compromised activities of daily life. This study is aimed to collect data regarding the functional status of patients due to vestibular and postural impairments with stroke. The study will be descriptive comparative cross-sectional. It will be conducted at Idress Hospital Sialkot. This study will be completed within the time duration of six months. Convenient sampling techniques will be used to collect the data. Both genders with equal ratio will be included in this study after fulfillments of inclusion and exclusion criteria. Visual vertigo analogue scale, Dix-Hallpike Maneuver, DHI (Dizziness Handicap Inventory), Posture assessment scale for stroke (PASS) score, Time up and go test will be used as data collection tools. All data will be collected after informed consent from patient. All data will be collected under complete supervision of physiotherapist. All the data will be demonstrated as mean and percentage. The analysis of data will be done by using SPSS.26(Statistical Package For social science) and Excel. Statistical significance will be set as P = 0.05. Frequency tables, pie charts, bar charts will be used to show summary of group measurements measured over time. Our analysis will provide the association of vestibular and postural impairments with functional status in both males and females after stroke

DETAILED DESCRIPTION:
Stroke (cerebrovascular accident CVA) is a medical condition associated with neurological deficits caused by interruption of blood flow to brain. Main types of strokes are ischemic (due to blood loss) and hemorrhagic (due to bleeding). Sign and symptoms of stroke may include inability to move or feel, problem understanding and speaking, dizziness, unable to walk and dependency in daily life. All these factors effect the functionality of the patient. If symptoms last less than one or two hours then it is transient ischemic stroke (TIA), also known as mini stroke. Modifiable risk factors associated with stroke are high blood pressure, smoking, diabetes, metabolic diseases and obesity. Male gender , ethnicity, family history , genetic predisposition and old age all are non-modifiable risk factors.

Vestibular dysfunction is define as the disturbance in body's balance system. It may be due to peripheral or central disorders. The peripheral cause for vestibular dysfunction is peripheral neuritis. The most common cause of the central vestibular dysfunction is an ischemic stroke of posterior fossa which contains brain stem and cerebellum. Vestibular dysfunction often present as dizziness. patients with vestibular dysfunction are at high risk of fall due to vertigo and gait imbalances, postural instability, increased sway and irregulated gate Risk factors associated with vestibular dysfunctions include female gender, age more than 40 years, depression and poor educational status.

The balance impairments in post stroke state is complex. It includes weight bearing asymmetry, muscles weakness, increased visual dependency and disturbed perceptions. All these factors effect the independent functionality of the patient. Postural instability increases after stroke which result in restriction in independence of daily activities.

There is relation between dizziness and stoke. Patients with dizziness or vertigo are at higher risk of stroke than general population. Dizziness is common in patients who experience stroke for the first time. Dizziness is a cognitive manifestation of disturbed balance system of body. Dizziness is a risk factor for fall and it has negative influence on quality of life.

Balance is defined as the ability to maintain the center of gravity within base of support with minimal postural sway. Balance is classified as static and dynamic balance. Static balance is associated with sitting and standing, while dynamic balance is associated with walking and running. Insufficient balance in stroke survivors due to sensory and motor deficits results in decrease activities of daily life and functional status.

Patients suffering from posterior inferior cerebral artery PICA stroke, present with vertigo, dizziness, vomiting, headache, gait changes, impairments in postural control and horizontal nystagmus ipsilateral to the lesion. These symptoms are result of a compromised vestibular afferent sensory input which impairs the motor output for the management/maintenance of balance.

The aim of this study is to find the association between vestibular and postural impairment on functional status of patients .Our study will also provide the difference of result between male and females whether they are equally effected or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-70
2. Male and female equal ratio
3. Mine-mental state examination (MMSE) more than 25
4. Confirmed ischemic stroke referred by neurologist using computerized tomography(CT)
5. Patient after 6 months of 1st ischemic stroke
6. Hypertensive patient

Exclusion Criteria:

1. Unstable cardiovascular status
2. Musculoskeletal conditions that influence posture e.g implants , orthodesis , fixation
3. Unable to follow verbal commands
4. Unable to keep any(sitting and standing) positions for 30 seconds.
5. Diabetic neuropathy

Ages: 35 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Vertigo Analogue Scale | Baseline (single reading)
  This scale indicates the amount of dzziness patient experince by covering distance of 10cm in different environments scoring 0-10.(43) The VVAS shows high validity and responsiveness to any change detected clinically. The VVAS can also be used to verify the progression of the client's symptoms.
Dix Hallpike Maneuver | Baseline (single reading)
  When performing the Dix-Hallpike test, patients are lowered quickly to a supine position (lying horizontally with the face and torso facing up) with the neck extended 30 degrees below horizontal by the clinician performing the maneuver
Diszziness Handicap Inventory | Baseline (single reading)
  The DHI is a 25-item self-report questionnaire that quantifies the impact of dizziness on daily life by measuring self-perceived handicap.
  Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0
.Posture assessment scale for stroke (PASS) score: | Baseline (single reading)
  it consist of 12 items which are assessed on 4 levels (0-3 points) on rating scale. It assesses the eligibility to maintain or change lying, sitting and standing posture.(46) This scale is easy to use and has good interrater and intra-rater reliability as well as internal consistency
Time up and go test | Baseline (single reading)
  * 10 seconds = normal ≤20 second = good mobility can go out alone, mobile without gait aid
  * 30 seconds = problems, cannot go outside alone, requires gait aid A score of ≥ 14 seconds has been shown to indicate high risk of falls

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan(Punjab_, Pakistan

IPD SHARING:
Plan to Share IPD: No